CLINICAL TRIAL: NCT03122561
Title: Estimation of Paracetamol in Urine to Assess the Diurnal Variation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BSMMU-013-CT
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Diurnal Variation of Paracetamol Excretion
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Healthy Volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paracetamol 500 mg tablet at Morning (Other): Urinary paracetamol of 41 healthy volunteers will be measured after oral administration at morning
  Interventions: Drug: Paracetamol 500 mg tablet at morning
- Paracetamol 500 mg tablet at Midday (Other): Urinary paracetamol of 41 healthy volunteers will be measured after oral administration at midday
  Interventions: Drug: Paracetamol 500 mg tablet at midday
- Paracetamol 500 mg tablet at Night (Other): Urinary paracetamol of 41 healthy volunteers will be measured after oral administration at night
  Interventions: Drug: Paracetamol 500 mg tablet at night

INTERVENTIONS:
Drug: Paracetamol 500 mg tablet at morning — Single dose oral paracetamol will be administered at 8.00 am
  Other Names: Tablet. Ace
  Arms: Paracetamol 500 mg tablet at Morning
Drug: Paracetamol 500 mg tablet at midday — Single dose oral paracetamol will be administered at 2.00 pm
  Other Names: Tablet. Ace
  Arms: Paracetamol 500 mg tablet at Midday
Drug: Paracetamol 500 mg tablet at night — Single dose oral paracetamol will be administered at 8.00 pm
  Other Names: Tablet. Ace
  Arms: Paracetamol 500 mg tablet at Night

SUMMARY:
Paracetamol is an antipyretic drug that is taken orally at different times of the day in same dose. It is excreted mainly through renal route which may show diurnal variation. In this study, urinary excretion of paracetamol of 41 healthy men of same age group will be measured by HPLC after oral administration of 500 mg paracetamol tablet at morning, midday and night. The measured values will be compared in order to adjust doses of oral paracetamol at different times of the day.

DETAILED DESCRIPTION:
Drug absorption, distribution, biotransformation and excretion are influenced by many different physiological functions of the body which may vary with time of the day. The time dependent changes in pharmacokinetics are due to circadian variation of human physiology and it is sometimes responsible for drug effects or adverse effects. Paracetamol is a widely used antipyretic and analgesic drug. It is usually well tolerated when used at the recommended dose. Paracetamol is a weak acidic drug that is rapidly absorbed and distributed after oral administration. It is metabolized extensively in liver and excrteted mainly through kidney as metabolites of paracetamol and some are as unchanged form. Paracetamol and its metabolites can be determined in biological fluids (urine, plasma, serum) by various mechanisms. High Performance Liquid Chromatography (HPLC) is a modern analytical chemistry technique by which paracetamol can be identified, separated and estimated from urine sample. This study is designed to investigate whether the excretion of paracetamol is changed or not if administered at same dose as oral tablet at three different times of the day. For this purpose after taking written informed consent 41 healthy men of aged 19- 23 will be provided 500 mg oral paracetamol tablet at morning, midday and night in two weeks interval and estimation of urinary paracetamol will be done by HPLC after paracetamol ingestion. A pilot study has been done and result shows highest concentration of paracetamol in urine after its oral administration found at 4th hour. Urine sample will be collected before and 4 hour after paracetamol administration in chloroform containing urine container and will be preserved in - 20 ̊C until analysis. Paracetamol standard has been collected from the same pharmaceutical company of which the drug will be used for study. Mobile phase will be consist of acetonitrile and distilled water and flow rate will be 0.5 ml/min at 25 ̊C temperature and 900 Psi pressure. The standard and sample will be analysed at a wavelength 254 nm. Total urinary paracetamol of that time will be estimated by multiplying total urinary volume in ml and concentration of paracetamol in one ml of urine. After measuring paracetamol at different times of the day, statistical analysis will be done to compare those values. If significant variation is found, adjustment of dose of oral paracetamol in different time of the day will be tried.

ELIGIBILITY:
Inclusion Criteria:

* The healthy male student volunteers of Eastern Medical College having age range between 19 and 23 years

Exclusion Criteria:

* Age <19 years , >23 years
* Volunteers on analgesic or antipyretic medication
* Volunteers with history of hypersensitivity to paracetamol
* Volunteers taking any enzyme inducing or enzyme inhibiting drug
* Volunteers with impaired renal or hepatic function

Ages: 19 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in the amount of urinary paracetamol in different times | [Morning: 0 hour (baseline), 4 hour (end); Mid-day: 0 hour (baseline), 4 hour (end); Night: 0 hour (baseline), 4 hour (end)] [Safety Issue: No]
  Changes in the amount of urinary paracetamol in different times (morning, midday and night) 4 hours after oral administration of 500 mg of paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, PhD, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Eastern Medical College, Comilla, Bangladesh

IPD SHARING:
Plan to Share IPD: No